CLINICAL TRIAL: NCT06738706
Title: Exploratory Study of the Impact of Intermittent Hypoxia-hyperoxia Training on Patients with Cerebral Venous Outflow Disorders
Brief Title: Intermittent Hypoxia-Hyperoxia Training in Cerebral Venous Outflow Disorders (IHHT-CVOD)
Acronym: IHHT-CVOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHHT-CVOD
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Venous Outflow Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent Hypoxia-Hyperoxia Training (Experimental): Participants will receive 14 times intermittent hypoxia-hyperoxia training interventions within 2 to 3 weeks.
  Interventions: Device: intermittent hypoxia-hyperoxia treatment

INTERVENTIONS:
Device: intermittent hypoxia-hyperoxia treatment — The intermittent hypoxia-hyperoxia training refers to 4 cycles of 10-minute hypoxia inhalation interspersed with 20-minute hyperoxia, which is performed once daily for 14 days within 2 to 3 weeks.

SUMMARY:
This study aims to investigate the safety and efficacy of intermittent hypoxia-hyperoxia treatment in patients with cerebral venous outflow disorders.

DETAILED DESCRIPTION:
Cerebral venous outflow disorder (CVOD), resulting from internal blockage, external oppression, or jugular valve incompetence, can cause hemodynamic disturbance and abnormal perfusion status. Restricted applicable populations and limited benefits constrain the application of existing CVOD management approaches. Previous studies indicate intermittent hypoxia hyperoxia training (IHHT) might improve circulatory status via hypoxic stimulation and allow hypoxic-related symptom amelioration through oxygen supply. Thus, IHHT might be a promising therapy for the CVOD population. Studies have so far proved inconclusive as to whether IHHT is safe and effective for CVOD. Therefore, the present study aimed to investigate the safety and feasibility of IHHT in patients with cerebral venous outflow disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 80 years.
2. Diagnosis of CVOD confirmed by CE-MRV, DSA, CTV, or ultrasound, including cerebral venous sinus stenosis (CVSS), internal jugular venous stenosis (IJVS), or internal jugular venous valve incompetence.
3. Unexplained chronic neurological deficits or other symptoms > 3 months.
4. Signed informed consent from the patient or legally authorized representative.

Exclusion Criteria:

1. Life-threatening comorbidities.
2. Clinical symptoms and signs explained by other diseases.
3. Intracranial hypertension; moderate to severe intracranial/extracranial arterial stenosis.
4. History of ischemic/hemorrhagic stroke or cerebral endovascular surgery.
5. Intracranial abnormalities, such as tumors, abscesses, vascular malformations, or cerebral venous sinus thrombosis.
6. Confirmed sleep apnea, plateau residency, traveling history of altitude > 1000m, or relative hypoxic exposure within last six months.
7. Poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | After the 14-time IHHT interventions.
  Adverse reactions included headache, vomiting, diarrhea, fatigue, dizziness, and insomnia.
Incidence of adverse reactions | After the first-time IHHT intervention.
  Adverse reactions included headache, vomiting, diarrhea, fatigue, dizziness, and insomnia.

SECONDARY OUTCOMES:
Heart rate | At the first-time IHHT intervention.
  Heart rate was recorded every 5 minutes from the start to 30 minutes following the completion of the first IHHT intervention.
Blood pressure | At the first-time IHHT intervention.
  Brachial arterial blood pressure was measured every 5 minutes from the start to 30 minutes following the completion of the first IHHT intervention.
Tissue oxygen saturation | At the first-time IHHT intervention.
  Peripheral and cerebral tissue oxygen saturations were recorded every 5 minutes from the start to 30 minutes following the completion of the first IHHT intervention.
Twenty-four-hour ambulatory blood pressure | The day before the 14-time treatment; The day after the 14-time treatment.
  Including systolic blood pressure and diastolic blood pressure (mmHg).
Blood routine indexes | The day before the 14-time treatment; The day after the 14-time treatment.
  Changes in blood routine indexes will be detected.
Blood biochemical changes | The day before the 14-time treatment; The day after the 14-time treatment.
  Changes in blood biochemical parameters will be detected.
The global impression of the treatment | The day after the 7-day treatment.
  The patient global impression of change (PGIC) scale was used after the 14 training sessions to assess the perceived global impression of change from the patient's perspective. This instrument is a numeric scale ranging from 1 (very much improved) to 7 (very much worse), with a lower score indicating better improvement.
Symptoms | The day before the 14-time treatment ;The day after the 14-time treatment.
  It is evaluated by completing the follow-up form.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No